CLINICAL TRIAL: NCT03656302
Title: Circadian Rhythm Dysregulation in Offspring of Parents With Bipolar Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Kowloon Hospital (Unknown); The Affiliated Hospital of Guangzhou Medical University (Guangzhou Huiai Hospital) (Unknown); Shenzhen Nanshan Center for Chronic Disease Control (Unknown); Shenzhen Baoan Center for Chronic Disease Control (Unknown); Shenzhen Longgang Center for Chronic Disease Control (Unknown); Shenzhen Futian Center for Chronic Disease Control (Unknown)
Responsible Party: Principal Investigator, Dr. Zhang Jihui, Assistant professor, Chinese University of Hong Kong
Other Study IDs: 03140636
Record Dates: First submitted 2018-07-05; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Circadian Rhythm Disorders; High-risk offspring; Endophenotypes
MeSH Terms: conditions — Bipolar Disorder; Chronobiology Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case offspring: Inclusion criteria:
  1) aged 6-21 years old; 2) having at least one biological parent with a lifetime or current diagnosis of bipolar disorder; 3) being able to read, write and understand Chinese; 4) both the offspring and her/his parent(s) agree to sign the informed consent form
  Exclusion criteria:
  1) having lifetime history or current diagnosis of bipolar disorder; 2) having no good ability to attend this project, such as patients with dementia and mental retardation.
- Control offspring: Inclusion criteria:
  1) aged 6-21 years old; 2) having no biological parent(s) with lifetime or current diagnosis of mood disorders. 3) being able to read, write and understand Chinese; 4) both the offspring and her/his parent(s) agree to sign the informed consent form.
  Exclusion criteria:
  1) having lifetime history or current diagnosis of bipolar disorder. 2) having no good ability to attend this project, such as patients with dementia and mental retardation.

SUMMARY:
This study aims to 1) investigate the differences and variances in circadian rhythms at several levels, including physical activity, dim light melatonin onset, diurnal patterns of cortisol, and body temperature between the offspring of patients with bipolar disorder (BD) and offspring of healthy parents by using a high-risk study design; and 2) determine whether these indicators correlate with psychopathological symptoms as measured by the psychometric measurements.

DETAILED DESCRIPTION:
Bipolar disorder (BD), characterized by episodes of mania or hypomania with frequent depressive episodes, is commonly found in the general population with a lifetime prevalence of 1-2% in the world. The morbidities and mortality associated with bipolar disorder are huge and the repercussion on their family members is considerate. Nonetheless, there is no existing well-established prevention strategy that may prevent this distressing mental disorder. A major reason is that there was limited understanding of the prodromal phase of BD. On the other hand, the genetic background determines about 60-85% of risk variance of BD. In other words, the offspring carries significant risk and propensity to develop future BD. Limited existing studies suggested that offspring of patients with BD have a higher rate of sleep and circadian disturbances and mental disorders than those offspring of parents without BD. Nonetheless, it is still unclear whether sleep and circadian disturbances are prodromal markers or risk factors for the development of bipolar disorder in this high-risk population.

In light of our research and other studies' preliminary findings on the relationship between circadian rhythms dysregulation and BD and robust heritability in BD, we hypothesize that

1. Circadian rhythm dysregulations are prodromal features and endophenotypes of BD. The offspring of BD parents will have more circadian rhythm dysregulations than those offspring of healthy controls;
2. The biologic indices of circadian rhythm dysregulations will be correlated with subsyndromal psychopathology.

ELIGIBILITY:
1. Case offspring

Inclusion criteria:

1) aged 6-21 years old; 2) having at least one biological parent with a lifetime or current diagnosis of bipolar disorder; 3) being able to read, write and understand Chinese; 4) both the offspring and her/his parent(s) agree to sign the informed consent form

Exclusion criteria:

1) having lifetime history or current diagnosis of bipolar disorder; 2) having no good ability to attend this project, such as patients with dementia and mental retardation.

2. Control offspring

Inclusion criteria:

1) aged 6-21 years old; 2) having no biological parent(s) with lifetime or current diagnosis of mood disorders. 3) being able to read, write and understand Chinese; 4) both the offspring and her/his parent(s) agree to sign the informed consent form.

Exclusion criteria:

1) having lifetime history or current diagnosis of bipolar disorder. 2) having no good ability to attend this project, such as patients with dementia and mental retardation.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with BD will be recruited from psychiatry outpatient clinics in Hong Kong and mainland China. Healthy parents will be recruited from our on-going community-based projects. In addition, the investigators will also recruit subjects through public advertisement through various media such as Facebook, poster, and emails. In view of the potential sex differences in these circadian rhythms indicators of interest, the adolescent offspring of healthy parents will be age- and sex-matched to the adolescent offspring of BD parents.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-02-11 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-06-28 (Estimated)

PRIMARY OUTCOMES:
Dim light melatonin onset (DLMO, free day) | 9 hours
  The subjects will be instructed to arrive at our sleep laboratory 9 hours before their usual bedtime. Saliva samples will be collected into clear sterile tubes every 30 minutes for eight hours, starting six hours before and 2 hours after individual's habitual bedtime. Subjects will be asked to stay in the light-controlled study room (<30 lux in any direction of gaze) and remain awake and sit quietly.

SECONDARY OUTCOMES:
Actigraphy and sleep diary | one week
  One-week Actigraphy (GENEActiv) and sleep diary will be employed to continuously measure sleep/wake patterns and physical activity.
Body temperature | one week
  Consecutive one-week period Skin temperature will be measured by iButton DS1921H (Dallas, Maxim) at 3 places: right on the middle of the frontal aspect of the thigh, abdomen (1 cm above the navel), and the right infraclavicular area. It has been demonstrated that iButton has satisfactory validity, reliability, and utility in the measurements of circadian rhythms and sleep/wake cycles.
Circadian rhythm pattern of salivary cortisol (free day) | 24 hours
  Subjects will be instructed to collect saliva samples using salivettes upon awakening (0 minute, 15 minutes, 30 minutes, and 45 minutes to measure cortisol awakening response) and then every 4 hours to measure the circadian rhythm patterns of cortisol secretion.
24-Hour Urinary 6-sulphatoxymelatonin (aMT6s) Assessment | 24 hours
  During the night of DLMO measure, all subjects will be instructed to collect a 24-h urinary samples (nearly 1000 mL) for the urinary 6-sulfatoxymelatonin assessment.
Sleep macroarchitecture by polysomnography | One-night (nearly 8 hours)
  One-night polysomnographic assessment will be measured to document the sleep architecture, together with DLMO measure. The recordings include electro-oculogram (EOG), electroencephalogram (EEG), electromyogram (EMG; monitoring over chin and bilateral anterior tibialis muscles), electrocardiogram (ECG), nasal-oral airflow and respiratory movements. The PSG data will be scored according to the most updated scoring manual of the American Academy of Sleep Medicine.
The rates of chronotype and sleep disorders | nearly one hour
  Chronotype will be estimated by the Morningness-eveningness Questionnaire (MEQ) or the Children's ChronoType Questionnaire (CCTQ). Sleep disorders, such as insomnia and delayed sleep phase disorder, will be also determined by the Diagnostic Interview for Sleep Patterns and Disorders (DISP).

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Zhang, PhD, Principal Investigator — Chinese University of Hong Kong; Yun Kwok Wing, MBChB, Study Chair — Chinese University of Hong Kong; Siu Ping Lam, Study Director — Shatin Hospital; Shirley Xin Li, PhD, Study Director — Hong Kong University; Roger Man Kin Ng, PhD, Study Director — Kowloon Hospital
Locations (1):
- Department of psychiatry, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lei B, Feng H, Yang L, Wang J, Chen J, Song W, Jiang C, Zhang K, Wang Q, Tsang JCC, Chan NY, Liu Y, Chan JWY, Pan J, Zhang B, Li T, Merikangas KR, Zhang J, Wing YK. Circadian rhythm dysfunction and psychopathology in the offspring of parents with bipolar disorder: a high-risk study in the Chinese population. Gen Psychiatr. 2024 May 22;37(3):e101239. doi: 10.1136/gpsych-2023-101239. eCollection 2024. PMID 38800632